CLINICAL TRIAL: NCT02523846
Title: Comparing Effectiveness of Post-operative Analgesia Between Patient Re-education and the Additional of a Basal Morphine Infusion to IV-PCA Morphine in Patients With Unsatisfactory Analgesia After Laparotomy
Brief Title: Patient Re-education vs. Background Morphine to IV-PCA in Patient With Unsatisfactory Analgesia Post Laparotomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinical Research Centre, Malaysia (Other)
Responsible Party: Principal Investigator, Yeoh Lee Choo, Anaesthesiologist, Clinical Research Centre, Malaysia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20790
Record Dates: First submitted 2015-08-10; First posted 2015-08-14 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-08

CONDITIONS: Post-operative Pain
Keywords: IV-Patient Controlled Analgesia (IV-PCA); background morphine infusion; patient re-education
MeSH Terms: conditions — Pain, Postoperative | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Background morphine infusion to IV-PCA Morphine (Active Comparator): Calculate based on patient's age, in mg/hour
  Interventions: Drug: morphine; Behavioral: Patient re-education
- Patient re-education to IV-PCA Morphine (Experimental): Using patient information leaflet
  Interventions: Behavioral: Patient re-education

INTERVENTIONS:
Drug: morphine — Investigators use the formula that was published by Pamela Macintyre in her paper entitled "Age is the Best Predictor of Postoperative Morphine Requirements." The estimation for the first 24-hour morphine requirement after surgery is calculated as: 100 - age (year).
  So, half of the total 24-hour morphine requirement will be infused over 24 hours.
  e.g. background morphine infusion= (100-Age)/ 2/ 24 (mg/hour)
  Arms: Background morphine infusion to IV-PCA Morphine
Behavioral: Patient re-education — A similar leaflet will be used to re-educate patient at 4 hour after surgery. The correct method to initiate IV-PCA dose, possible side effects and addiction issue will be explained again and re-emphasized

SUMMARY:
The purpose of this study is to improve IV-Patient Controlled Analgesia (IV-PCA) technique for postoperative analgesia. Investigators are comparing between patient re-education and the background morphine infusion among patients who fail to achieve satisfactory analgesia using IV-PCA Morphine after laparotomy.

DETAILED DESCRIPTION:
In this study, investigators have a second inclusion criteria for subject recruitment. For subjects who meet this criteria meaning their dynamic pain (when blowing incentive spirometer) is ≥ 4/10 after starting on IV-PCA Morphine will be randomized in to 2 groups. One group will receive patient re--education with an additional background morphine infusion and the other group will receive re--education only.

The second highlight for this study is regarding the background morphine calculation. The background morphine is calculated according to this formula:

Total morphine requirement in the first 24 hours post surgery (mg) = 100 - Age (year) So, the background morphine infusion will be calculated based on subject's age and half of their 24 hours requirement will be infused over 24 hours.

This formula was published by Pamela Macintyre in her paper titled " Age is the Best Predictor of Postoperative Morphine Requirement".

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA)Physical Status Classification Class I and II
* Elective laparotomy
* able to understand either malaysia, mandarin, english language or local dialect
* patient with dynamic pain score 4/10 and more within the first 4-hour after initiation of IV-PCA

Exclusion Criteria:

* patient refusal
* laparotomy with pfannenstiel incision
* patients with a history of allergy to opioids
* patients who required post-operative ventilation support
* patients ASA III and above
* patients unable to use PCA due to insufficient comprehension
* morbid obesity/ obstructive sleep apnea
* chronic opioid or alcohol abuse

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
measure pain intensity at rest and when blowing incentive spirometer (dynamic pain) | 48 hours after surgery
  use combination of Numerical Rating Scale(NRS) and Visual Analogue Scale(VAS)

SECONDARY OUTCOMES:
respiratory rate | 48 hours after surgery
total accumulative morphine consumption from IV-PCA pump | 48 hours after surgery
sedation level | 48 hours after surgery
  sedation score (0 to 3)

CONTACTS AND LOCATIONS:
Overall Officials: lee choo yeoh, master, Principal Investigator — CRC Malaysia
Locations (1):
- Sultanah Bahiyah Hospital, Alor Seatr, Kedah, Malaysia

REFERENCES:
- [Result] Macintyre PE, Jarvis DA. Age is the best predictor of postoperative morphine requirements. Pain. 1996 Feb;64(2):357-364. doi: 10.1016/0304-3959(95)00128-X. PMID 8740614